CLINICAL TRIAL: NCT00849979
Title: M.D. Anderson Symptom Inventory (MDASI-GI) Validation and Clinical Utility in Patients With Gastrointestinal Cancers Being Treated or Followed by GI Medical Oncology
Brief Title: Validating M.D. Anderson Symptom Inventory (MDASI-GI) in GI Cancer Patients Under Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2007-0228
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Gastrointestinal Cancer
Keywords: Colorectal; Gastric; Gastrointestinal; GI; Liver; Pancreas; Gastrointestinal Cancers; Gastro-Intestinal Chemotherapy; M.D. Anderson Symptom Inventory; MDASI-GI; Medical Oncology
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Questionnaire (Other)
  Interventions: Behavioral: Questionnaire
- Questionnaire + Interview (Other)
  Interventions: Behavioral: Questionnaire; Other: Interview

INTERVENTIONS:
Behavioral: Questionnaire — Day 1 MDASI-GI Questionnaire
Other: Interview — Open-ended, audiotaped interviews
  Arms: Questionnaire + Interview

SUMMARY:
The goal of this study is to learn more about the symptoms that may occur in patients with GI cancer. The types of GI cancer being studied are cancers of the stomach, liver, pancreas, colon, and rectum. Researchers want to test a newly-designed questionnaire called the M. D. Anderson Symptom Inventory - Gastrointestinal (MDASI-GI) questionnaire.

DETAILED DESCRIPTION:
Questionnaires:

If you agree to take part in this study, you will be asked to complete the MDASI-GI questionnaire on Day 1. It asks about any symptoms you may be experiencing, and how those symptoms may be interfering with your daily life. You will also complete two questionnaires that ask about the overall quality of your life. In total, these questionnaires should take about 20 minutes to complete.

You will then complete a questionnaire that asks for demographic information such as your age and marital status. It should take about 5 minutes.

You will receive another copy of the MDAS-GI questionnaire and the quality-of-life questionnaire to take home and complete 1 week later. The research staff will call you to remind you when it is time to complete this questionnaires. You should mail it back to the study staff in a stamped, pre-addressed envelope that will be provided to you.

Evaluation of Questionnaires:

Also on Day 1, a small group of participants (25 out of the 185 total participants) will complete an additional questionnaire called a "cognitive debriefing" questionnaire. These 25 participants will be the first 5 participants to join this study who have 1 of the 5 types of cancer being studied.

The questionnaire asks questions related to how easy it was for you to answer the questions on the MDASI-GI questionnaire, whether the questions relate to the symptoms you may be experiencing, and whether any other questions should be added. This questionnaire should take about 10 minutes to complete.

Interview:

Another small group of participants (a different 25 out of the 185 total) will have a one-on-one interview with a member of the study staff. During the interview, you will be asked to further describe the symptoms you may have experienced. This interview will be scheduled for a day when you are going to be at M. D. Anderson for a routine clinic visit. It should take about 30 minutes to complete.

You and the interviewer will be the only ones in the room during the interview, and the information collected will be kept confidential. The interview will be tape-recorded.

Questionnaire and Interview Content:

Your responses will not be shared with your doctor. If you feel you need a doctor's opinion about anything that is asked about, please contact your doctor.

Information Collection:

As part of this research study, the research staff will collect information from your medical record one time. This will include data about the cancer, cancer treatment, and routine test results.

Length of Study Participation:

After you mail back the questionnaire at Week 1 (or complete it by phone interview with research staff), or after the interview if you have one, your active participation in this study will be over.

This is an investigational study. Up to 185 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be out-patients being reviewed or treated in M. D. Anderson's Department of GI Medical Oncology.
* Patients will have received a confirmed pathological diagnosis of GI cancer (gastric cancer, liver cancer, pancreatic cancer, colorectal cancer).
* Patients will or will not be undergoing chemotherapy or treatment with other agents on the day of enrollment.
* Patients must be > or = 18 years of age.
* Patients must be able to speak and read English.

Exclusion Criteria:

* Patients who, in research staff's estimation, cannot understand the intent of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Validation of M. D. Anderson Symptom Inventory - Gastrointestinal (MDASI-GI) Questionnaire (Response) | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Xin Shelley Wang, MD, MPH, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org